CLINICAL TRIAL: NCT04931875
Title: Total-body 18F-FDG PET / CT in the Evaluation of Treatment and Prognosis of Patients With Lymphoma
Brief Title: Total-body PET / CT in the Evaluation of Treatment and Prognosis of Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Yumei Chen, deputy head of the department of nuclear medicine, RenJi Hospital
Other Study IDs: KY2021-052
Record Dates: First submitted 2021-06-15; First posted 2021-06-18 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Lymphoma
Keywords: Lymphoma, Total-body PET/CT, Prognosis, Dynamic Imaging
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Total-body PET/CT (uExplorer): The diagnostic value of dynamic parameters(K1、Ki etc) to evaluate the prognosis of lymphoma compared to the static ones(SUV、MTV、TLG etc).
  Interventions: Device: Total body PET/CT (uExplorer)

INTERVENTIONS:
Device: Total body PET/CT (uExplorer) — A total-body PET/CT scanner (uEXPLORER) with a 194-cm scan range will be applied in patients affected with lymphoma.

SUMMARY:
The prospective study aims to explore the value of total-body PET/CT dynamic imaging (uExplorer) in assessing the treatments and prognosis in patients affected with lymphoma. Total-body 18F-FDG PET/CT scans are being performed before treatment, after three cycles of chemotherapy and six weeks after the end of treatment. The plan of this study involves to evaluate the clinical application of total-body PET / CT in patients histopathologically-diagnosed as lymphoma, and to optimize the dynamic acquisition protocols with total-body 18F-FDG PET/CT.

DETAILED DESCRIPTION:
100 cases of lymphoma patients are enrolled in this study. Participation in this study involves three dynamic 18F-FDG PET/CT exams, which occur before the treatments start, two or three days before the fourth cycle of chemotherapy, and then six weeks after the end of last treatments. Progress Free Survival(PFS) and Overall Survival(OS) are used as the end points to study the value of metabolic parameters obtained from the dynamic PET/CT imaging. The differences of dynamic metabolic parameters and static SUV value are evaluated in patients with lymphoma from the perspective of diagnosis, staging, treatment and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated informed consent prior to any study specific procedures
* Had histologically confirmed lymphoma
* Patients aged 18~75 years old

Exclusion Criteria:

* Female patients who are pregnant, breast-feeding
* Currently active second malignancy other than Lymphoma
* Any situation not suitable for this study judged by researchers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients with lymphoma will be scanned by total-body 18F-FDG uEXPLORER PET/CT
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2023-05-20 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
PFS | three years after last patient recruited
  Progress-free survival is calculated from the date of randomization to the date of the first progress at any site or death from any cause or censored at the date of the last follow-up.
OS | three years after last patient recruited
  The duration from the date of random assignment to the date of death from any cause or censored at the date of the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Yumei Chen, Ph.D;M.D., Principal Investigator — RenJi Hospital
Locations (1):
- Shanghai jiaotong University School of Medicine, Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen Y, Zhou M, Liu J, Huang G. Prognostic Value of Bone Marrow FDG Uptake Pattern of PET/CT in Newly Diagnosed Diffuse Large B-cell Lymphoma. J Cancer. 2018 Mar 14;9(7):1231-1238. doi: 10.7150/jca.23714. eCollection 2018. PMID 29675104
- [Background] Zhou M, Chen Y, Liu J, Huang G. A predicting model of bone marrow malignant infiltration in 18F-FDG PET/CT images with increased diffuse bone marrow FDG uptake. J Cancer. 2018 Apr 19;9(10):1737-1744. doi: 10.7150/jca.24836. eCollection 2018. PMID 29805699
- [Background] Zhang X, Cherry SR, Xie Z, Shi H, Badawi RD, Qi J. Subsecond total-body imaging using ultrasensitive positron emission tomography. Proc Natl Acad Sci U S A. 2020 Feb 4;117(5):2265-2267. doi: 10.1073/pnas.1917379117. Epub 2020 Jan 21. PMID 31964808
- [Background] Zhang YQ, Hu PC, Wu RZ, Gu YS, Chen SG, Yu HJ, Wang XQ, Song J, Shi HC. The image quality, lesion detectability, and acquisition time of 18F-FDG total-body PET/CT in oncological patients. Eur J Nucl Med Mol Imaging. 2020 Oct;47(11):2507-2515. doi: 10.1007/s00259-020-04823-w. Epub 2020 May 18. PMID 32424483
- [Background] Zhou M, Chen Y, Huang H, Zhou X, Liu J, Huang G. Prognostic value of total lesion glycolysis of baseline 18F-fluorodeoxyglucose positron emission tomography/computed tomography in diffuse large B-cell lymphoma. Oncotarget. 2016 Dec 13;7(50):83544-83553. doi: 10.18632/oncotarget.13180. PMID 27835875